CLINICAL TRIAL: NCT07213700
Title: The International Registry for Alzheimer's Disease and Other Dementias (InRAD): An International Registry Observational Study Dedicated to Evaluating Outcomes Data in Alzheimer's Disease
Brief Title: InRAD Observational Study
Acronym: InRAD
Status: Not yet recruiting | Type: Observational
Sponsor: Stichting International Registry for Alzheimer's Disease and other Dementias Foundation (Other)
Collaborators: InRAD Foundation (Data Processor) (Unknown); All Individual Principal Investigators and their centers (Data Controllers) (Unknown)
Responsible Party: Sponsor
Other Study IDs: InRAD-AD-OBS-V1.0
Record Dates: First submitted 2025-09-23; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease(AD); Mild Cognitive Impairment (MCI); Subjective Cognitive Decline (SCD); Non-Alzheimer Degenerative Dementia
Keywords: Alzheimer's disease (AD); Dementia; Observational study; Real-world data (RWD); International registry; Cognitive decline; Lecanemab; InRAD Registry; InRAD Foundation; Cognitive screening (MoCA, MMSE); AD-specific therapies; Clinical staging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer's Disease Registry Participants: Individuals diagnosed with Alzheimer's disease or undergoing diagnostic work-up, enrolled in the InRAD Registry for long-term observational follow-up. This cohort includes treated, treatment-eligible, and untreated patients across global clinical centers participating in routine care and data collection.
  Interventions: Other: None, this is a non-interventional observational study

INTERVENTIONS:
Other: None, this is a non-interventional observational study — None applicable

SUMMARY:
The goal of this international observational study is to evaluate long-term disease outcomes and treatment safety in people with Alzheimer's disease (PwAD), by collecting real-world data from routine clinical practice across global clinical centers.

The InRAD Registry Observational Study has several aims:

* To collect medical information for many years from a large group of people with Alzheimer's disease. This will be used for research, which will support improved understanding about the disease.
* To enable researchers to look at the effectiveness, usefulness and safety of treatments for Alzheimer's disease.
* To enable researchers to answer similar research questions and compare results in many different areas of the world.

People with Alzheimer's disease who meet the eligibility criteria and agree to participate in the Study will be asked to visit their doctor (e.g. psychiatrist, geriatrician, or neurologist) at least once a year, or as frequently as is needed for their care. During or after their appointments they may be offered assessments, tests, medications, and treatments as determined by their doctor and their team. This is an observational data collection.

DETAILED DESCRIPTION:
The study protocol is owned by all InRAD Observational Study Investigators. All centers taking part in InRAD are the data controllers. InRAD is a data processor and is providing operational management and system support.

Study Type: Prospective, non-interventional, multinational observational cohort study.

Study Objective: The primary goal of the InRAD Observational Study is to collect and analyze real-world data (RWD) to evaluate long-term disease outcomes and treatment safety in people with Alzheimer's disease (PwAD). The study aims to:

* Assess disease stage transitions, cognitive and functional changes over time.
* Examine the relationship between demographics, comorbidities, diagnostic and monitoring tests, drug exposures, and outcomes.
* Compare disease demographics and outcomes across countries and regions.
* Characterize the occurrence of medical events, including Serious Adverse Events (SAEs) and Adverse Events (AEs), particularly in relation to AD-specific treatments.

Study Population: Adults undergoing diagnostic work-up for Alzheimer's disease or already diagnosed. Includes treated, treatment-eligible, and untreated patients. Participants must be attending an InRAD Center and provide informed consent for long-term follow-up.

Recruitment and Consent: Recruitment is open to global clinical centers with qualified investigators. Informed consent is obtained from patients and, where applicable, their caregivers. Consent includes authorization to share pseudonymized demographic and medical data with the InRAD Registry.

Data Collection: Investigators use the InRAD Web cloud-based data-entry platform and agree to collect the defined Minimum Dataset at least annually for their patients:

Minimum Dataset (MDS):

* Patient demographics
* Disease characteristics
* Clinical outcomes
* Safety data
* Treatment details

In addition to the Minimum Dataset, Investigators may collect a variety of disease-specific or other data-fields of interest from the Extended Dataset:

Extended Dataset (EDS):

* Lifestyle factors
* Biomarkers and imaging data
* Care partner information
* Quality of life and burden assessments

Centers, through their PIs, and the InRAD SLG (Scientific Leadership Group), may propose research analyses and cohort sub-studies of interest to be conducted using the pooled Registry dataset or subsets of the Registry data.

For each analysis and sub-study proposal, the Center, through its PI, always exclusively decide whether to participate and contribute their Center data for use in the research.

The IT tool is owned, maintained and freely provided by the InRAD Foundation to Member Centers to enable and support the Study.

Pseudonymized data is to be submitted to the InRAD registry at least biannually and may be updated more frequently depending on clinical practice.

Governance and Oversight: The study is coordinated by the InRAD Foundation and governed by its Scientific Leadership Group (SLG). Each participating center is responsible for obtaining Ethics Committee (EC) or Institutional Review Board (IRB) approval unless exempt. No Data Monitoring Committee (DMC) is appointed, consistent with the non-interventional nature of the study.

Safety Monitoring: SAEs and other medical events are recorded using MedDRA coding. Centers are responsible for reporting SAEs to local authorities and manufacturers. The registry supports longitudinal safety analyses to identify treatment-related risks.

Participant Reimbursement: No financial reimbursement is provided. Diagnostic and treatment costs are covered by patients, their healthcare provider or their health insurance.

Sampling: The study does not use randomization or stratified sampling. Instead, it includes all eligible and consenting patients encountered during routine care at participating centers, reflecting a real-world clinical population.

Funding: InRAD is coordinated by the independent International Registry for Alzheimer's Disease and Other Dementias Foundation, a health-related not-for-profit entity incorporated in the Netherlands.

InRAD has received financial contributions from the pharmaceutical industry. InRAD does not endorse any companies or products. InRAD is operated independently from these companies.

ELIGIBILITY:
Inclusion Criteria:

* Be undergoing diagnostic work-up for Alzheimer's disease (AD), OR
* Have a confirmed diagnosis of AD (whether currently treated with an AD-specific treatment, or untreated),
* Be attending an InRAD Center,
* Have provided informed consent for long-term follow-up

Exclusion Criteria:

-Any patient or legal representative who is unable or unwilling to provide a signed informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be from centers part of the InRAD international network
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2036-01 (Estimated); Study Completion 2036-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Alzheimer's Disease Clinical Staging over time | 10 years
  Use of the "Clinical staging for individuals on the Alzheimer's disease continuum" NIA-AA 2018/24 criteria, ranging from Stage 0 to Stage 6:
  * Stage 0 Asymptomatic, deterministic gene;
  * Stage 1 Asymptomatic, biomarker evidence only;
  * Stage 2 Transitional decline: mild detectable change, but minimal impact on daily function;
  * Stage 3 Cognitive impairment with early functional impact;
  * Stage 4 Dementia with mild functional impairment;
  * Stage 5 Dementia with moderate functional impairment;
  * Stage 6 Dementia with severe functional impairment.

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized individual participant data (IPD) collected through the InRAD data entry system will be shared with InRAD investigators/researchers. Shared IPD will include data from the MDS (minimum data set) and EDS (extended data set)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 1 year after international deployment of the registry platform
Access Criteria: Access to IPD is granted to qualified researchers affiliated with participating InRAD Centers. Data requests must be submitted via the InRAD Registry platform and approved by the Scientific Leadership Group (SLG). Approved researchers will receive encrypted, pseudonymized datasets under a Data Use Agreement that ensures confidentiality, secure handling, and deletion after the permitted access period.

REFERENCES:
- [Background] Perneczky R, Darby D, Frisoni GB, Hyde R, Iwatsubo T, Mummery CJ, Park KH, van Beek J, van der Flier WM, Jessen F. Real-world datasets for the International Registry for Alzheimer's Disease and Other Dementias (InRAD) and other registries: An international consensus. J Prev Alzheimers Dis. 2025 Apr;12(4):100096. doi: 10.1016/j.tjpad.2025.100096. Epub 2025 Feb 18. PMID 39971671
- See also: InRAD Foundation website — https://www.inradnetwork.org/